CLINICAL TRIAL: NCT02321007
Title: Study of Placental Function in Healthy and Pathological Pregnancies
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1073
Record Dates: First submitted 2014-12-03; First posted 2014-12-19 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to establish a tissue and data repository consisting of samples of human placentas, umbilical cord blood, and maternal blood, collected at the time of delivery. Specimens will be used in cellular, molecular, and functional studies to learn more about changes in placental structure and function, which can result in serious pregnancy complications and determine life-long health by programming the fetus for future metabolic and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women delivering at term
* Women with pregnancy complications such as:

  * pre-term birth,
  * intrauterine growth restriction,
  * diabetes, and
  * obesity.

Exclusion Criteria:

* Women:

  * under stress,
  * experiencing pain of labor.
* Pregnancies complicated by other pathologies.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women delivering at term as well as women with pregnancy complications such as pre-term birth, intrauterine growth restriction, diabetes and obesity will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2014-09; Primary Completion 2031-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Collecting, processing, and archiving human specimens from 1250 subjects | Specimens will be stored for 50 years in repository
  Human placental tissue, umbilical cord blood, and maternal blood samples will be collected from pregnant women at the time of their delivery. The samples will be used to enhance understanding of the role of the placenta in the development of pregnancy complications and in programming of adult disease.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jansson, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No